CLINICAL TRIAL: NCT00604630
Title: German Multicenter EPO Stroke Trial (Phase II/III)
Brief Title: Multicenter Efficacy Study of Recombinant Human Erythropoietin in Acute Ischemic Stroke
Acronym: ESS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Max-Planck-Institute of Experimental Medicine (Other)
Collaborators: Johnson & Johnson (Industry); Parexel (Industry)
Responsible Party: Prof. Dr. Dr. Hannelore Ehrenreich (MD, DVM), Head of the Division of Clinical Neuroscience, Max-Planck-Institute of Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BfArM-4019639/2002; "EPO Stroke Study"; "Ehrenreich EPO Stroke Study"; "Ehrenreich Study"
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-09

CONDITIONS: Infarction, Middle Cerebral Artery; Middle Cerebral Artery Stroke; Stroke, Acute
Keywords: stroke; EPO; erythropoietin; ischemia; hypoxia; antiapoptosis; neuroprotection; rtPA; thrombolysis; stroke, middle cerebral artery; Ischemic stroke in the middle cerebral artery territory
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Stroke; Ischemia; Hypoxia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): 50ml 0.9% NaCL
  Interventions: Drug: 0.9% NaCl
- verum (Active Comparator): erythropoietin alfa 40,000 IU iv in 50ml 0.9% NaCl
  Interventions: Drug: recombinant human erythropoietin alfa

INTERVENTIONS:
Drug: recombinant human erythropoietin alfa — 40,000 IU in 50ml 0.9% NaCl iv on 3 consecutive days, starting within 6 hours after onset of symptoms
  Other Names: ERYPO
  Arms: verum
Drug: 0.9% NaCl — 50ml 0.9% NaCl iv on 3 consecutive days, starting within 6 hours after onset of symptoms
  Arms: placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled multicenter study is to determine in a cohort of 506 patients with acute ischemic stroke in the middle cerebral artery territory, the effect of a three-day high-dose, intravenous erythropoietin treatment on functional outcome up to a follow-up of 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke in the middle cerebral artery territory
* Clearly defined time of onset
* Confirmed by MRI (DWI, Flair)
* NIH Stroke Scale ≥ 5
* Age > 18 years
* Treatment within 6h after onset of symptoms
* Informed consent by patient, relatives or independent physician
* Life expectancy > 90 days

Exclusion Criteria:

* Coma or precoma (level of consciousness ≥ 2 in NIH Stroke Scale)
* Previous stroke within the same territory
* Intracranial or subarachnoidal hemorrhage
* Traumatic brain injury or brain operation within the last 4 weeks
* Neoplasia, septic embolism, infectious endocarditis
* MRI contraindications
* Renal failure (i.e. dependent on dialysis)
* Known malignant/life-threatening disease
* Known myeloproliferative disorder, polycythemia
* Known allergy or antibodies against erythropoietin
* Participation in other intervention trials
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2003-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Neurological/functional outcome as measured by the Barthel Index (BI) | day 90

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) responder | day 90
Barthel Index (BI) | day 30
mRS | day30, day 90
NIH Stroke Scale | day 1, 3, 7, 30, 90
Proportion of subjects with minimal disability (mRS 0-1) | day 30, day 90
All-cause mortality | day 90
Mortality directly related to stroke | day 90
Proportion of subjects with BI >= 95 | day 30, day 90
Proportion of subjects with BI=100 | day 30, day 90
Proportion of subjects with neurological recovery | day 3, 7, 30, 90
Distribution of mRS scores | day 30, day 90
Distribution of BI scores | day 30, day 90
Distribution of NIH Stroke Scale scores | day 30, day 90
Serum level of glial damage markers S100B and GFAP | day 1, 2, 3, 4, 7
Lesion size (MRI DWI, flair) | day 1, day 7
Overall survival | day 90
Late recovery index (BI day 90 versus BI day 30) | day 30 to day 90

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (9):
  - Neurologische Klinik des Städtischen Klinikums Braunschweig, Braunschweig
  - Neurologische Klink, Klinikum Bremen-Mitte, Bremen
  - Neurologische Klinik, Allgemeines Krankenhaus Celle, Celle
  - Klinik und Poliklinik für Neurologie, Universitätsklinikum Carl Gustav Carus der TU Dresden, Dresden
  - Neurologische Klinik, Universität Erlangen-Nürnberg, Erlangen
  - Klinik für Neurologie, Universität Essen, Essen
  - Neurologische Universitätsklinik der Georg-August-Universität Goettingen, Göttingen
  - Neurologische Klinik, Medizinische Hochschule Hannover, Hanover
  - Klinik und Poliklinik für Neurologie der Universität Leipzig, Leipzig

REFERENCES:
- [Background] Siren AL, Fratelli M, Brines M, Goemans C, Casagrande S, Lewczuk P, Keenan S, Gleiter C, Pasquali C, Capobianco A, Mennini T, Heumann R, Cerami A, Ehrenreich H, Ghezzi P. Erythropoietin prevents neuronal apoptosis after cerebral ischemia and metabolic stress. Proc Natl Acad Sci U S A. 2001 Mar 27;98(7):4044-9. doi: 10.1073/pnas.051606598. Epub 2001 Mar 20. PMID 11259643
- [Background] Ehrenreich H, Hasselblatt M, Dembowski C, Cepek L, Lewczuk P, Stiefel M, Rustenbeck HH, Breiter N, Jacob S, Knerlich F, Bohn M, Poser W, Ruther E, Kochen M, Gefeller O, Gleiter C, Wessel TC, De Ryck M, Itri L, Prange H, Cerami A, Brines M, Siren AL. Erythropoietin therapy for acute stroke is both safe and beneficial. Mol Med. 2002 Aug;8(8):495-505. PMID 12435860
- [Background] Lewczuk P, Hasselblatt M, Kamrowski-Kruck H, Heyer A, Unzicker C, Siren AL, Ehrenreich H. Survival of hippocampal neurons in culture upon hypoxia: effect of erythropoietin. Neuroreport. 2000 Nov 9;11(16):3485-8. doi: 10.1097/00001756-200011090-00017. PMID 11095504
- [Background] Siren AL, Knerlich F, Poser W, Gleiter CH, Bruck W, Ehrenreich H. Erythropoietin and erythropoietin receptor in human ischemic/hypoxic brain. Acta Neuropathol. 2001 Mar;101(3):271-6. doi: 10.1007/s004010000297. PMID 11307627
- [Background] Herrmann M, Ehrenreich H. Brain derived proteins as markers of acute stroke: their relation to pathophysiology, outcome prediction and neuroprotective drug monitoring. Restor Neurol Neurosci. 2003;21(3-4):177-90. PMID 14530580
- [Background] Ehrenreich H, Hasselblatt M, Knerlich F, von Ahsen N, Jacob S, Sperling S, Woldt H, Vehmeyer K, Nave KA, Siren AL. A hematopoietic growth factor, thrombopoietin, has a proapoptotic role in the brain. Proc Natl Acad Sci U S A. 2005 Jan 18;102(3):862-7. doi: 10.1073/pnas.0406008102. Epub 2005 Jan 10. PMID 15642952
- [Background] Siren AL, Radyushkin K, Boretius S, Kammer D, Riechers CC, Natt O, Sargin D, Watanabe T, Sperling S, Michaelis T, Price J, Meyer B, Frahm J, Ehrenreich H. Global brain atrophy after unilateral parietal lesion and its prevention by erythropoietin. Brain. 2006 Feb;129(Pt 2):480-9. doi: 10.1093/brain/awh703. Epub 2005 Dec 9. PMID 16339796
- [Background] Ehrenreich H, Hinze-Selch D, Stawicki S, Aust C, Knolle-Veentjer S, Wilms S, Heinz G, Erdag S, Jahn H, Degner D, Ritzen M, Mohr A, Wagner M, Schneider U, Bohn M, Huber M, Czernik A, Pollmacher T, Maier W, Siren AL, Klosterkotter J, Falkai P, Ruther E, Aldenhoff JB, Krampe H. Improvement of cognitive functions in chronic schizophrenic patients by recombinant human erythropoietin. Mol Psychiatry. 2007 Feb;12(2):206-20. doi: 10.1038/sj.mp.4001907. Epub 2006 Oct 10. PMID 17033631
- [Background] Ehrenreich H, Fischer B, Norra C, Schellenberger F, Stender N, Stiefel M, Siren AL, Paulus W, Nave KA, Gold R, Bartels C. Exploring recombinant human erythropoietin in chronic progressive multiple sclerosis. Brain. 2007 Oct;130(Pt 10):2577-88. doi: 10.1093/brain/awm203. Epub 2007 Aug 29. PMID 17728357
- [Derived] Woywodt A, Gerdes S, Ahl B, Erdbruegger U, Haubitz M, Weissenborn K. Circulating endothelial cells and stroke: influence of stroke subtypes and changes during the course of disease. J Stroke Cerebrovasc Dis. 2012 Aug;21(6):452-8. doi: 10.1016/j.jstrokecerebrovasdis.2010.11.003. PMID 21852153
- [Derived] Ehrenreich H, Weissenborn K, Prange H, Schneider D, Weimar C, Wartenberg K, Schellinger PD, Bohn M, Becker H, Wegrzyn M, Jahnig P, Herrmann M, Knauth M, Bahr M, Heide W, Wagner A, Schwab S, Reichmann H, Schwendemann G, Dengler R, Kastrup A, Bartels C; EPO Stroke Trial Group. Recombinant human erythropoietin in the treatment of acute ischemic stroke. Stroke. 2009 Dec;40(12):e647-56. doi: 10.1161/STROKEAHA.109.564872. Epub 2009 Oct 15. PMID 19834012
- See also: homepage of the Max-Planck-Institute of Experimental Medicine — http://www.em.mpg.de